CLINICAL TRIAL: NCT04212520
Title: Predictive Value of Non-fasting Blood Lipid Levels for Cardiovascular and Cerebrovascular Events in Community Population(PICC Study)
Brief Title: Predictive Value of Non-fasting Blood Lipid Levels for Cardiovascular Events in Community Population(PICC Study)
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018150H(R2)
Record Dates: First submitted 2019-12-24; First posted 2019-12-27 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Lipid
Keywords: non-fasting lipid; cardiovascular and cerebrovascular events; major adverse cardiovascular events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study will collect 20 mL whole blood samples from subjects at one or more study visits. The whole blood will be processed to plasma and stored for testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Numerous studies have shown that non-fasting blood lipid levels are closely related to the occurrence of cardiovascular and cerebrovascular events, but it is still unclear in the Chinese population. The purpose of the study is to investigate the association between non-fasting blood lipid levels and adverse outcomes in Chinese community population.

DETAILED DESCRIPTION:
Study population includes subjects who living in community, of any race or ethnicity, 18 or older years of age, and have provided written informed consent to provide biological sample at one or more study visits. Physical examination, questionnaire survey and biological sample collection will be conducted at baseline and the incidence of a composite of major adverse cardiovascular events will be investigated during follow-up.

ELIGIBILITY:
Inclusion Criteria:

•≥18 years old;

* Signed informed consent;
* Life expectancy is greater than 1 year.

Exclusion Criteria:

* mental disorder;
* is not willing to participate in the clinical study;
* suffered with other disease to quite the trial;
* violated the protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population includes subjects who living in community, of any race or ethnicity, 18 or older years of age, and have provided written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Through study completion, an average of 1 years
  All-cause mortality was confirmed through a combination of hospital medical records, telephone contacts with patients or family members, and death registration at the Center for Disease Control and Prevention.
Cardiovascular Mortality | Through study completion, an average of 1 years
  Cardiovascular mortality was defined as death attributable to an ischemic cardiovascular cause (including fatal cardiovascular events and stroke).
Cardiovascular and cerebrovascular diseases | Through study completion, an average of 1 years
  The number of and the incidence rate of cardiovascular and cerebrovascular diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ying-qing, PhD, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China